CLINICAL TRIAL: NCT00005027
Title: A Phase II Study of Rebeccamycin Analog in Renal Cell Cancer
Brief Title: Rebeccamycin Analog in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067548; U01CA062487 (NIH); P30CA022453 (NIH); WSU-C-2063; NCI-T99-0113
Record Dates: First submitted 2000-04-06; First posted 2003-08-08 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — becatecarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: becatecarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of rebeccamycin analog in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with advanced renal cell carcinoma when treated with rebeccamycin analogue.
* Assess the quantitative and qualitative toxicities associated with this drug in this patient population.

OUTLINE: Patients receive rebeccamycin analogue IV over 30-60 minutes daily for 5 days. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 23-44 patients will be accrued for this study within 9-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced unresectable, locally recurrent, or metastatic renal cell carcinoma not eligible for a higher priority trial
* Measurable disease

  * Longest diameter at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan
* No nonmeasurable disease only including:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses not confirmed and followed by imaging techniques
  * Cystic lesions
* No known brain metastases

  * History of brain metastases that have been resected and/or irradiated with subsequent normal brain CT scan allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of any site
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to rebeccamycin analogue
* No other concurrent uncontrolled illness (e.g., ongoing or active infection)
* No concurrent psychiatric illness or social situation that would preclude study compliance
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed
* Recovered from toxic effects

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics

Other:

* No other concurrent investigational or commercial agents or therapies for renal cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Ibrahim D, Hussain M, LoRusso P, et al.: Rebeccamycin analog (BMY-27557-14) in renal cell cancer (RCC): preliminary results of a phase II trial. [Abstract] Proceedings of the American Society of Clinical Oncology A-2373, 2001.